CLINICAL TRIAL: NCT03807232
Title: Predictive Factors, Demographics and Mortality for ARDS in Burn Patients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: ARDS in Burn Patients USZ
Record Dates: First submitted 2018-09-13; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: ARDS, Human; Burns; Lung Diseases
Keywords: ARDS, Human; Burns; Lung Diseases; Risk Factors; Retrospective Studies; Decision Support Techniques
MeSH Terms: conditions — Respiratory Distress Syndrome; Burns; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pbARDS: Burn patients who developed post-burn ARDS
- No pbARDS: Burn patients without development of post-burn ARDS

SUMMARY:
This retrospective study characterizes the clinical course and identifies four independent predictors of Acute Respiratory Distress Syndrome (ARDS) after burn injury (post-burn ARDS; pbARDS). In addition, a clinically useful prognostic score for pbARDS is introduced (ARDS burn score), which was derived from these independent predictors. The newly developed score may be helpful for the development of specific treatment strategies.

DETAILED DESCRIPTION:
Rationale:

Acute Respiratory Distress Syndrome (ARDS) after burn injury (post-burn ARDS; pbARDS) is a severe complication associated with a mortality of up to 44%. To date, only few studies have been published on the clinical course and predictive factors of pbARDS.

Objectives:

To characterize the clinical course of pbARDS, to identify relevant predictors, including the development of a prognostic score, and to examine outcome parameters such as mortality and hospitalization days.

Methods:

A retrospective analysis of 400 patients admitted to the Burns Intensive Care Unit of the University Hospital Zurich from 2004 to 2009 was performed. Multivariate logistic regression was used to determine independent risk factors for pbARDS. A prognostic score was developed, which was tested with leave-one-out-cross-validation and Receiver Operating Characteristic (ROC) curves.

ELIGIBILITY:
Inclusion Criteria:

all patients treated at the Burns Intensive Care Unit (BICU) of the University Hospital Zurich (USZ) between January 2004 and December 2009.

Exclusion Criteria:

Exclusions were made because of incomplete or unavailable data, re-hospitalization due to complications of previous burns, and the initial decision not to resuscitate due to unfavorable prognosis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated at the Burns Intensive Care Unit (BICU) of the University Hospital Zurich (USZ) between January 2004 and December 2009
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-08-26 (Actual); Primary Completion 2013-05-23 (Actual); Study Completion 2013-05-23 (Actual)

PRIMARY OUTCOMES:
Incidence of post-burn ARDS | 6 years
  Number of patients who developed post-burn ARDS among 400 Patients admitted to Burns Intensive Care Unit of University Hospital Zurich
Clinical course of post-burn-ARDS | 6 years
  various clinical parameters related to the Outcome of post-burn-ARDS
predictors of post-burn ARDS | 6 years
  To identify relevant predictors of post-burn ARDS, including the development of a prognostic score

SECONDARY OUTCOMES:
to examine outcome parameter mortality | 6 years
  A retrospective analysis of 400 patients admitted to the Burns Intensive Care Unit of the University Hospital Zurich
to examine outcome parameter hospital stay | 6 years
  A retrospective analysis of 400 patients admitted to the Burns Intensive Care Unit of the University Hospital Zurich

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Giovanoli, Prof. Dr. med., Study Chair — Universitätsspital Zürich

IPD SHARING:
Plan to Share IPD: No